CLINICAL TRIAL: NCT04422652
Title: Combination of Novel Therapies for CKD Comorbid Depression (CONCORD)
Brief Title: Combination of Novel Therapies for CKD Comorbid Depression
Acronym: CONCORD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Susan Hedayati, MD, PROFESSOR, IM-Nephrology, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-2020-0046; R01DK124379 (NIH)
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Diseases; Major Depressive Disorder; End Stage Kidney Disease (ESRD)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Depressive Disorder, Major; Kidney Failure, Chronic | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Those eligible will be randomized via a computerized random number generator 1:1:1 to BAT, bupropion, or control, using block randomization, stratified by site and CKD stage (3b, 4, 5-non dialysis, and 5-dialysis). Randomization assignment will be obtained via the secure web portal hosted at UTSW. As in previous trials that involve therapy for MDD, it is challenging to double-blind aspects of this study that involve BAT. However, we have made every effort to maintain blind as much as possible. Bupropion for Strategy 2 and double-blind matching placebo for the control arm will be administered by concealed allocation. Participants in Strategy 1 will receive matching placebo by single-blind allocation. Although it is impossible to conceal the allocation of the BAT to the research team, it is intended for the participants to remain single-blinded to BAT vs. CM. Using Computer Assisted Telephone Interviewing, the same assessor, blinded to interventions, will assess outcomes for both sites.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Strategy 1 (Active Comparator): Strategy 1: Single-blind Behavioral Activation Therapy plus placebo for 8 weeks (Phase 1), augmented in non-remitters at 8 weeks with single-blind bupropion (Phase 2) for another 8 weeks.
  Interventions: Behavioral: Behavioral activation therapy; Drug: Placebo
- Strategy 2 (Active Comparator): Strategy 2: Double-blind bupropion plus single-blind Clinical Management (CM) attention control for 8 weeks (Phase 1), augmented in non-remitters at 8 weeks with single-blind BAT (Phase 2) for another 8 weeks.
  Interventions: Drug: Bupropion; Other: Clinical Management
- Control (Placebo Comparator): Control: Clinical management attention control plus placebo for 16 weeks
  Interventions: Drug: Placebo; Other: Clinical Management

INTERVENTIONS:
Drug: Bupropion — Bupropion is an anti-depressant medication.
  Other Names: Wellbutrin
  Arms: Strategy 2
Behavioral: Behavioral activation therapy — Brief behavioral activation treatments administered via video tele-conferencing.
  Arms: Strategy 1
Drug: Placebo — Double-blind placebo.
  Arms: Control; Strategy 1
Other: Clinical Management — Clinical management will serve as the attention control for the Behavioral Activation Therapy intervention.
  Arms: Control; Strategy 2

SUMMARY:
The overall goal of the study is to determine if treatment of a Major Depressive Disorder (MDD) improves the outcomes of patients with chronic kidney disease (CKD). We showed that MDD is present in 25% of CKD patients and independently associated with progression to End-Stage Kidney Disease, hospitalization, and death. Depression is also associated with lower quality of life (QOL), fatigue, poor sleep, and non-adherence to diet and medications. However, evidence for efficacy and tolerability of commonly-used antidepressant medications or nonpharmacologic treatments are limited in CKD patients. Our group was the first to conduct a double-blind randomized controlled trial for MDD treatment in 201 patients with non-dialysis CKD, and showed that sertraline, a commonly used selective serotonin reuptake inhibitor (SSRI), was no more efficacious than placebo for improving depressive symptoms. It becomes imperative to test novel strategies to treat MDD in CKD. We propose to compare with a control group, the efficacy and tolerability of two novel treatment strategies - (1) Behavioral Activation Teletherapy (BAT) for 16 weeks, with the addition of bupropion, a non-SSRI antidepressant, at 8 weeks for patients whose depression has not remitted (non-remitters); and (2) bupropion for 16 weeks, with the addition of BAT at 8 weeks for non-remitters. In Aim 1, we will investigate the efficacy and tolerability of these 2 strategies vs. control for improvement in a primary endpoint of depressive symptoms in 201 patients (67 per group) with CKD stages 3b-5 and MDD at 2 sites, randomized 1:1:1 to either strategy or a control group of Clinical Management plus placebo. We hypothesize that either approach vs. control will result in a minimal clinically important difference of 2 points improvement in depressive symptoms, as ascertained blindly by the Quick Inventory of Depressive Symptomatology. In Aim 2 we will investigate the efficacy and tolerability of 8 weeks of (1) single-blind BAT plus placebo or (2) double-blind bupropion plus Clinical Management vs. control for improvement in depressive symptoms. In Aim 3, we will compare the efficacy of these 2 treatments strategies vs. control for improvement in CKD patient-centered outcomes including a. adherence to medications and healthcare visits; b. fatigue; c. sleep; and d. overall functioning. A clinical trial is urgently needed to address the evidence gap that exists for MDD treatment in CKD patients.

DETAILED DESCRIPTION:
Aim 1. Compare the efficacy and tolerability of two 16-week strategies vs. control for treatment of CKD patients with MDD starting with (1) BAT or (2) bupropion, each augmented to a combination of both in non-remitters. Primary hypothesis: Treatment with either strategy will improve depression (primary endpoint) and be tolerable.

Patients with stages 3b-5 CKD and MDD (N=201) will be randomized 1:1:1 to 16 weeks of:

Strategy 1: Single-blind BAT plus placebo, augmented in non-remitters at 8 weeks with single-blind bupropion; Strategy 2: Double-blind bupropion plus single-blind Clinical Management (CM) attention control, augmented in non-remitters at 8 weeks with single-blind BAT; Control: CM attention control plus placebo. There will be >80% power to detect a minimal clinically important difference (MCID) of 2 points on the Quick Inventory of Depressive Symptomatology between each intervention and control, assuming a 14% attrition rate.

Exploratory aim (a): Explore if remote access to therapy via internet vs. travel to clinic affects treatment efficacy.

Aim 2. Investigate efficacy and tolerability of 8 weeks (Phase 1) of (1) BAT plus placebo or (2) bupropion plus CM, vs. control, for improvement in depression. Secondary hypothesis: Treatment with 8 weeks of BAT or bupropion will improve depression. There will be 80% power to detect a MCID of 2 points between each arm and control, assuming 10% attrition.

Exploratory aims:

(a) Investigate whether patient preference for BAT vs. drug affects treatment efficacy; (b) compare efficacy of each combination in Phase 2 with control; (c) compare change from baseline in plasma C-reactive protein in drug vs. BAT or control arms.

Aim 3. Investigate the efficacy of these two 16-week treatment strategies vs. control for improvement in CKD patient-centered outcomes including: (a) adherence to medications and healthcare visits; (b) fatigue; (c) sleep; (d) overall functioning. Secondary hypothesis: Treatment with either strategy will result in clinically meaningful improvements in adherence, fatigue, sleep and overall functioning in patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults aged 18 years or greater. There will be no upper age limit.
2. Presence of CKD stages 3b, 4 or 5, with an estimated glomerular filtration rate (GFR) of <45 mL/min/1.73 m2 for a period of at least 3 months, as defined by the National Kidney Foundation and determined using the four-variable Modification of Diet for Renal Diseases Study formula.
3. Presence of a current Major Depressive Disorder (MDD) based on MINI DSM IV-based criteria
4. Quick Inventory of Depressive Symptomatology-Self-report (QIDS-SR) score of ≥11 at enrollment and ≥11 on QIDS-Clinician Rated (QIDS-C) at randomization.
5. Able to understand and sign informed consent after the nature of the study has been fully explained
6. Kidney transplant patients that are at least 6 month post-transplantation (3 months post-transplant, with at least another 3 months to confirm eGFR <45)

Exclusion Criteria:

1. Unable to understand or give informed consent.
2. Unwilling or unable to participate in the protocol or comply with any of its components
3. Significant hepatic dysfunction or liver enzyme abnormalities 3 times or greater than the upper limit of normal
4. Terminal chronic obstructive pulmonary disease or cancer
5. Presence of seizure disorder
6. Current use of class I anti-arrhythmic medications (such as 1C propafenone and flecanide), pimozide, MAO inhibitors, reserpine, guanethidine, cimetidine, or methyldopa; tri-cyclic anti-depressants, neuroleptics, or anti-convulsants
7. Use of serotonergic drugs or supplements such as triptans, tramadol, linezolid, tryptophan, and St. John's Wort.
8. Use of medications known to cause QT prolongation on EKG
9. Ongoing use of antidepressant medications for depression treatment
10. Past treatment failure on bupropion
11. Initiation of depression-focused psychotherapy in the 3 months prior to study entry
12. Active alcohol or substance abuse or dependence that requires acute detoxification at study entry
13. Present or past psychosis or Bipolar I or II disorder
14. Dementia or a Mini-Mental State Examination score <23
15. Active suicidal intent
16. Pregnancy, lactation, or women of childbearing potential not willing to use adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology-Clinician Rated scale (QIDS-C) | Assessed at baseline and weeks 4, 6, 8, 12, and 16
  Assess the change from baseline in the QIDS-C total score in each of the intervention arms vs. the control arm. The score on the QIDS-C ranges from 0-27, with higher scores indicating more severe depressive symptoms.

SECONDARY OUTCOMES:
Serious adverse events | Assessed at weeks 4, 6, 8, 12, and 16.
  Pre-specified serious adverse events include death, hospitalization, renal replacement therapy (dialysis or kidney transplantation), and acute suicidal intent.
Quick Inventory of Depressive Symptomatology-Clinician Rated scale (QIDS-C) | Assessed at baseline and weeks 4, 6, and 8.
  Assess the change from baseline in the QIDS-C total score in each of the intervention arms vs. the control arm during the first 8 weeks of the study when participants in the treatment arms will be receiving monotherapy with BAT or bupropion.
Serious adverse events with monotherapy | Assessed at weeks 4, 6, and 8.
  Pre-specified serious adverse events include death, hospitalization, renal replacement therapy (dialysis or kidney transplantation), and acute suicidal intent during the first 8 weeks of the study.
Quick Inventory of Depressive Symptomatology-Clinician Rated scale (QIDS-C) | Assessed at weeks 8, 12, and 16.
  Assess the change from baseline in the QIDS-C total score in each of the intervention arms vs. the control arm during the second 8 weeks of the study when participants who did not respond to the treatment arms will be receiving combination therapy with BAT and bupropion.
High sensitivity C-reactive protein | Assessed at baseline and week 8
  Change from baseline to Week 8 in the plasma level of high sensitivity C-reactive protein (hsCRP) in the intervention groups vs. control.
Adherence to medications by Pill Count | Assessed at weeks 4, 8, 12, and 16.
  The proportion of participants in each arm that are adherent to antidepressant medications (or placebo, prescribed in the setting of the clinical trial). Adherence will be defined as 80% or greater of study drug taken.
Fatigue assessed by the Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) scale | Assessed at baseline and weeks 4, 8, 12, and 16
  Change from baseline in the FACIT-F scale in the intervention groups vs. control. The FACIT has 13 items, each on a Likert scale, with a score range of 0-52, and higher scores indicating a lower level of fatigue.
Sleep assessed by the Insomnia Severity Index (ISI) | Assessed at baseline and weeks 4, 8, 12, and 16
  Change from baseline in the Insomnia Severity Index (ISI) in the intervention groups vs. control. The ISI has 7 items that measure insomnia severity, with higher scores indicating more severe insomnia.
Overall functioning assessed by the Sheehan Disability Scale (SDS) | Assessed at baseline and weeks 4, 8, 12, and 16
  Change from baseline in the SDS in the intervention groups vs. control groups. The SDS assesses functional impairment in 3 domains: work, social life, and family, each evaluated on a 10-point visual analog scale, which are summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired).

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hedayati, MD, Principal Investigator — Stony Brook University
Locations (4):
- United States (4):
  - Stony Brook University Medical Center, Stony Brook, New York
  - Parkland Health and Hospital System, Dallas, Texas
  - UT Southwestern and Affiliates, Dallas, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Briggs LC. Hominid evolution in Northwest Africa and the question of the North African "Neanderthaloids". Am J Phys Anthropol. 1968 Nov;29(3):377-85. doi: 10.1002/ajpa.1330290312. No abstract available. PMID 5710375